CLINICAL TRIAL: NCT03835338
Title: WATCHMAN for Concomitant Left Atrial Appendage Electrical Isolation and Occlusion to Treat Persistent Atrial Fibrillation Rhythm
Acronym: WATCH-Rhythm
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor discretion
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2236
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Intervention Model Description: Treatment Arm - PVI, LAA Isolation and WATCHMAN LAAC Implantation Control Arm - PVI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test Group (Experimental): The test group will receive Pulmonary Vein Isolation, LAA Isolation and LAA Occlusion with the WATCHMAN LAAC Device
  Interventions: Device: Pulmonary Vein Isolation; Device: LAA Isolation; Device: LAA Occlusion
- Control Group (Active Comparator): The control group will receive Pulmonary Vein Isolation
  Interventions: Device: Pulmonary Vein Isolation

INTERVENTIONS:
Device: Pulmonary Vein Isolation — Pulmonary Vein Isolation by RF Ablation
Device: LAA Isolation — LAA Isolation by RF Ablation
  Arms: Test Group
Device: LAA Occlusion — LAA Occlusion by implantation of the WATCHMAN LAAC Device
  Arms: Test Group

SUMMARY:
WATCH-Rhythm is a prospective, randomized, multi-center, investigation to collect safety and effectiveness data on combining conventional AF ablation with LAA electric isolation and closure within a single procedure.

DETAILED DESCRIPTION:
WATCH-Rhythm is a prospective, randomized, multi-center, investigation to collect safety and effectiveness data on combining conventional AF ablation with LAA electric isolation and occlusion within a single procedure.

The primary objective is to test the effectiveness of adding LAA electrical isolation and closure to conventional atrial fibrillation versus conventional atrial fibrillation alone in treating patient with persistent atrial fibrillation from a single procedure.

This study will be conducted at up to 10 global sites in the European Union (United Kingdom, Spain, Germany, or others). The maximum enrollment ceiling for the Watch-Rhythm study is 278 subjects. Included in the enrollment ceiling are up to 20 roll-in subjects and a maximum of 258 randomized subjects.

The duration of the study is expected to last approximately 4 years. Enrollment is expected to take approximately 24 months. The duration of individual subject participation is expected to last approximately 2 years but may vary per subject.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is of legal age to participate in the study per the laws of their respective geography.
2. The subject has documented non-valvular persistent AF. For this protocol, the definition of persistent AF is sustained arrhythmia lasting at least 7-days but less than 36 months.
3. The subject is able to tolerate OAC post ablation.
4. Subject is able to undergo TEE.
5. The subject or legal representative is able to understand and willing to provide written informed consent to participate in the trial
6. The subject is willing and capable of attending all follow-up visits at the investigational site as medically appropriate.

Exclusion Criteria:

1. The subject is unable or unwilling to return for required follow-up visits and examinations.
2. The subject had or is planning to have any invasive cardiac procedure within 30 days prior to randomization (e.g., cardioversion, ablation).
3. Previous AF ablation (surgical or percutaneous).
4. Prior MAZE procedure.

4. The subject is planning to have any cardiac or non-cardiac invasive or surgical procedure that would necessitate stopping or modifying the protocol required medication regimen within 90 days after the WATCHMAN Closure Device implant (e.g., cardioversion, ablation, cataract surgery).

5. The subject had a prior BARC type 3 or 4 bleeding event within the 14 days prior to randomization. Lack of resolution of related clinical sequelae, or planned and pending interventions to resolve bleeding/bleeding source, are a further exclusion regardless of timing of the bleeding event.

6. The subject had a prior stroke (of any cause) or TIA within the 30 days prior to randomization.

7. The subject had a prior BARC type 3 or 4 bleeding event within the 14 days prior to randomization. Lack of resolution of related clinical sequelae, or planned and pending interventions to resolve bleeding/bleeding source, or a further exclusion regardless of timing of the bleeding event.

8. The subject has a history of atrial septal repair or has an ASD/PFO device. 9. The subject has an implanted mechanical valve prosthesis in any position. 10. The subject suffers from New York Heart Association Class IV Congestive Heart Failure.

11. Subject has LVEF <30% 12. Subject has hypertrophic cardiomyopathy. 13. The subject has had a myocardial infarction (MI) documented in the clinical record as either a non-ST elevation MI (NSTEMI) or as an ST elevation MI (STEMI), with or without intervention, within 90 days prior to randomization.

14. The subject is of childbearing potential and is, or plans to become pregnant during the time of the study (method of assessment upon study physician's discretion).

15. The subject is currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility.

16. The subject has a documented life expectancy of less than two years. 17. The subject has a known or suspected hypercoagulable state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from AF | 12 months
  Not having any of the following after the blanking period:
  * a documented symptomatic AF event (episode of 30 sec duration or longer by Holter, event monitor or rhythm strip; or for the full 10 second recording of a standard 12 lead ECG)
  * treatment with a Class I or Class III AAD
  * a documented symptomatic AF event (episode of 30 sec duration or longer by Holter, event monitor or rhythm strip; or for the full 10 second recording of a standard 12 lead ECG)
  * treatment with a Class I or Class III AAD